CLINICAL TRIAL: NCT03678870
Title: Discharge Opioid Education to Decrease Opioid Use After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Osmundson, Assistant Professor, Ob/Gyn, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181190
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Opioid Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Opioid Education
  Interventions: Other: Opioid Education Handout
- Control (No Intervention): standard discharge instructions, which lists medications prescribed at discharge

INTERVENTIONS:
Other: Opioid Education Handout — a single page handout with information about how to use medications for pain after discharge.
  Arms: Education

SUMMARY:
Background: The number of opioid overdose deaths in the United States has quadrupled in 15 years, a dramatic manifestation of the current opioid abuse epidemic. This rise parallels a sharp increase in the amount of legal prescription opioids dispensed. The abundance of prescription opioids available is a primary pathway for opioid abuse and diversion and higher opioid use after surgery has been associated with an increased risk of chronic opioid use. Reducing the amount of opioid used after cesarean delivery may decrease the risk of chronic opioid use and will help towards better estimating and reducing the amount of opioids prescribed at discharge.

Objective: To to compare discharge opioid education to standard care to ascertain whether opioid education reduces opioid use after hospital discharge

DETAILED DESCRIPTION:
Background: The number of opioid overdose deaths in the United States has quadrupled in 15 years, a dramatic manifestation of the current opioid abuse epidemic. This rise parallels a sharp increase in the amount of legal prescription opioids dispensed. The abundance of prescription opioids available is a primary pathway for opioid abuse and diversion and higher opioid use after surgery has been associated with an increased risk of chronic opioid use. Reducing the amount of opioid used after cesarean delivery may decrease the risk of chronic opioid use and will help towards better estimating and reducing the amount of opioids prescribed at discharge.

Objective: To to compare discharge opioid education to standard care to ascertain whether opioid education reduces opioid use after hospital discharge

Preliminary Data: Our soon to be published study (Obstetrics & Gynecology Journal) found that 30% of women used all their opioids after discharge for cesarean delivery because they "were following directions" and not because they had pain.

Enrollment & Randomization

Enrollment

* Participants will be approached after their cesarean delivery either in the recovery room or in their private postpartum room
* Informed written consent will be obtained by a trained research assistant (i.e. medical student) or by the study researchers (Attendings, fellows)
* After enrollment, participants will be asked to complete Survey 1 either in person or by giving sending them the web link with RedCap

Randomization

* Enrolled patients will be randomized in a 1:1 ratio using permuted blocks of 6
* Randomization sequence will be developed through sealed envelope.com
* Randomization and allocation will be done through RedCap

Study Procedures

1. Enrollment
2. Postoperative Day 0-1: Survey 1 through RedCap (takes ~10 minutes)
3. Randomization education versus usual care

   1. Control = Standard discharge instructions, which list medications prescribed at discharge
   2. Intervention = a single page handout (see attachment) with information about how to use medications for pain after discharge. This handout contains the following instructions

      * Get baseline pain control with ibuprofen
      * Use your opioid prescription only if your pain is very bad
      * Taper your medications
      * Get rid of leftover opioid tablets
4. At discharge all patients will receive the follow medications using PillsyCaps. These are standard medications given at discharge at our institution

   * Ibuprofen 600mg: 30 tablets
   * Hydrocodone 5mg -acetaminophen 325mg: 30 tablets
5. Postoperative day 14: All participants will be contacted to complete Survey 2 (Takes ~ 15 minutes

   * Attempts to contact each participant will be done 3 times before they are designated as "lost to follow up"
   * If a participant is still using opioids on postoperative day 14, they should be contacted weekly until they are no longer taking opioids

Primary Outcome Median number of tablets of hydrocodone-acetaminophen used after hospital discharge

Secondary Outcomes:

* Visual Analog Scale pain score (median)
* Percentage of patients reporting pain since discharge as worse than expected
* Percentage of patients obtaining additional prescriptions for pain
* Percentage of patients with unscheduled visits for pain
* Mean ibuprofen milligrams used hours 24-47 after cesarean
* Mean acetaminophen milligrams used hours 24-47 after cesarean
* Total Morphine Milligram Equivalents (MME) used per hour of inpatient stay

Risks

o Breach of confidentiality of protected health information

Reporting Adverse Events Any adverse events or unanticipated problems involving risk to participants or others will be reported to the Institutional Review Board and the Vanderbilt University Medical Center (VUMC) privacy office within 7 days of discovery.

Study Withdrawal/discontinuation Participants may withdraw at any time by providing written intent to the Primary Investigator. Participants may be removed from the study if they develop a major surgical complication after their cesarean.

Statistical Considerations

Using prior data, the average opioid MME used per person was 130 MME (SD 90) in the "average use" group. With an alpha of 5% and a beta of 80%, we estimate that 160 total participants are required to show a 30% reduction in opioid used. Assuming a lost to follow up rate of 20%, we plan to enroll 200 women.

Follow-up and Record Retention On average 100 cesareans are performed per month. With a 50% enrollment rate, we anticipate this study will take 4 months to complete

The patient list will be destroyed upon data analysis and publication. Redcap will be archived upon publication.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years old
* Women undergoing cesarean delivery at VUMC

Exclusion Criteria:

* Major post-surgical complications:
* cesarean hysterectomy, bowel or bladder injury, reoperation, ICU admission, wound infection or separation
* Chronic opioid use: Taking buprenorphine during pregnancy, taking an opioid for > 7 days during pregnancy.
* Women who do not speak English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women undergoing cesarean delivery at VUMC
Enrollment: 196 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Osmundson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Sarah Osmundson, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schirle LM, Dietrich MS, Lam L, Stone AL, Bruehl S, Osmundson SS. Accuracy of patient-reported versus real-time electronic postoperative opioid use outcomes. Am J Obstet Gynecol MFM. 2021 Jul;3(4):100347. doi: 10.1016/j.ajogmf.2021.100347. Epub 2021 Mar 11. No abstract available. PMID 33716134
- [Derived] Lam L, Richardson MG, Zhao Z, Thampy M, Ha L, Osmundson SS. Enhanced discharge counseling to reduce outpatient opioid use after cesarean delivery: a randomized clinical trial. Am J Obstet Gynecol MFM. 2021 Jan;3(1):100286. doi: 10.1016/j.ajogmf.2020.100286. Epub 2020 Dec 3. PMID 33451618

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education | Control
Started | 97 | 99
Completed | 84 | 91
Not Completed | 13 | 8
Not completed — prescribed non- protocol medications | 10 | 6
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education | Control | Total
Number analyzed (Participants) | 84 | 91 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.4) | 30.5 (4.9) | 30.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 91 | 175
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 52 | 60 | 112
  African-American | 20 | 15 | 35
  Other | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 84 | 91 | 175
High school education or less [Count of Participants; unit: Participants] — Women who completed high school (12th grade) or less
  Participants | 14 | 23 | 37

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use
Description: Median number of tablets of hydrocodone-acetaminophen used after hospital discharge
Time Frame: 6 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: hydrocodone tablets
Arm/Group | Education | Control
Number analyzed (Participants) | 84 | 91
hydrocodone tablets | 7.5 [2 to 15] | 10 [2 to 16]

2. Secondary Outcome: Disposed of Opioids Correctly
Description: Frequency of women reporting that they either returned their unused opioids to a pharmacy or flushed them down the toilet
Time Frame: 6 weeks postpartum
Population: Denominator includes only women who had leftover opioids
Measure: Number; unit: participants
Arm/Group | Education | Control
Number analyzed (Participants) | 79 | 83
participants | 30 | 14

3. Secondary Outcome: Analgesic Quiz Score
Description: Median score on an assessment of characteristics of analgesics including side effects, risks, and benefits. Score 1-10 for each question. Higher score is better.
Time Frame: 6 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education | Control
Number analyzed (Participants) | 84 | 91
score on a scale | 10 [9 to 10] | 8 [7 to 9]

4. Secondary Outcome: Additional Prescriptions
Description: Percentage of patients obtaining additional prescriptions for pain
Time Frame: 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Education | Control
Number analyzed (Participants) | 84 | 91
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Education | Control
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/99
Other Adverse Events (participants affected / at risk) | 0/97 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03678870/Prot_SAP_000.pdf